CLINICAL TRIAL: NCT03922282
Title: A Prospective, Randomized, and Controlled Study of the Safety and Efficacy in Gasless BABA(Bilateral Axillo-breast Approach) Robotic Thyroidectomy
Brief Title: BABA Robotic Thyroidectomy Without Gas is Safe Enough as That Use a Gas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Dongsik Bae, Assistant Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-08-009-004
Record Dates: First submitted 2019-02-20; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Thyroidectomy; Thyroid Diseases
Keywords: Gasless; Bilateral axillo-breast approach; Da Vinci; Robot-assisted thyroid surgery
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gasless BABA (Experimental): BABA robotic-thyroidectomy that do not using carbon dioxide but using elevation of flap.
  Interventions: Procedure: Gasless BABA
- Classic BABA (Active Comparator): BABA robotic-thyroidectomy using carbon dioxide.
  Interventions: Procedure: Classic BABA

INTERVENTIONS:
Procedure: Gasless BABA — BABA robotic-thyroidectomy that is using elevation of flap instead of using carbon dioxide.
  Arms: Gasless BABA
Procedure: Classic BABA — BABA robotic-thyroidectomy that is using carbon dioxide.
  Arms: Classic BABA

SUMMARY:
In this study, a randomized controlled study was conducted between two groups of 14 classic recipients of Carbon dioxide insufflation during BABA robotic-thyroidectomy and 14 recipients of Gasless method during BABA robotic-thyroidectomy. This is a study to see if there is any difference in hemodynamic and metabolic changes and pain .

ELIGIBILITY:
Inclusion Criteria:

* Subject who will have thyroid surgery

Exclusion Criteria:

* Subject who underwent thyroid surgery
* Subject who underwent any radiotherapy on neck
* Subject who need to neck dissection
* Subject under 18 years or over 70 years
* Bad general condition
* High American Society of Anesthesiologists(ASA) score (over 3)
* Breast feeder or pregnancy
* Subject who disagree to do this trial

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
heart rate | Change from baseline heart rate at the end of surgery
  heart rate in beats per minute
mean arterial pressure | Change from baseline mean arterial pressure at the end of surgery
  mean arterial pressure in mmHg
cardiac index | Change from baseline cardiac index at the end of surgery
  cardiac index in L/min/m^2, divide the cardiac output by the person's body surface area, measured by the Vigileo monitor, normal range is 2.5 to 4.5L/min/m2
cardiac output | Change from baseline cardiac output at the end of surgery
  cardiac output in L/minute, calculated by multiplying the stroke volume by the heart rate, measured by the Vigileo monitor
pH | Change from baseline pH at the end of surgery
  pH
PaCO2 | Change from baseline PaCO2 at the end of surgery
  PaCO2 in mmHg
VAS(visual analog score) | change from baseline VAS up to 3days after surgery
  Visual Analog Score for pain, range from 0 to 10, Higher the values represents more pains
BHC(bottom hit count) | change from baseline BHC up to 3days after surgery
  bottom hit count from intravenous patient controlled analgesia for pain
number of analgesics | change from baseline number of analgesics up to 3days after surgery
  number of analgesics(additional ketorolac uses)

CONTACTS AND LOCATIONS:
Locations (1):
- Dong sik Bae, Busan, South Korea